CLINICAL TRIAL: NCT05638126
Title: A Phase I Single and Multiple Ascending Dose and Food Effect Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HRS-1780 Tablets in Healthy Male Subjects
Brief Title: Safety and Tolerance of Increased Doses of HRS-1780 Tablets in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS-1780-101
Record Dates: First submitted 2022-11-24; First posted 2022-12-06 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2022-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): HRS-1780 table or placebo single dose
  Interventions: Drug: HRS-1780 table or placebo
- Part 2 (Experimental): HRS-1780 table or placebo single dose with food effect
  Interventions: Drug: HRS-1780 table or placebo
- Part 3 (Experimental): HRS-1780 table or placebo multiple dose
  Interventions: Drug: HRS-1780 table or placebo

INTERVENTIONS:
Drug: HRS-1780 table or placebo — HRS-1780 table or placebo single dose
  Arms: Part 1
Drug: HRS-1780 table or placebo — HRS-1780 table or placebo single dose with food effect
  Arms: Part 2
Drug: HRS-1780 table or placebo — HRS-1780 table or placebo multiple dose
  Arms: Part 3

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I clinical study. The primary objective is to evaluate the safety, tolerability, PK, and PD of single- and multiple-dose HRS-1780 in healthy subjects, and to evaluate the food effect on PK of HRS-1780.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years old (including boundary value, whichever is at the time of signing the informed consent form), healthy male.
2. Weight ≥50 kg, body mass index (BMI = body mass/height square (kg/m2)) is in the range of 18-28 (including boundary values)
3. Obtain informed consent before any activity related to the experiment begins, have a full understanding of the purpose and significance of the experiment, and be willing to comply with the test plan and dietary requirements.
4. Subjects (including partners) have no family planning within 3 months from the beginning of the signing of the informed consent form to the last dose, and are willing to adopt the efficient contraceptive measures stipulated in the program and guarantee not to donate sperm.

Exclusion Criteria:

1. People with a history of hypertension.
2. People with severe systemic infectious diseases, serious trauma or major surgical surgery before screening; those who plan to undergo surgery during the trial
3. There has been a history of clinical abnormal gastric emptying and severe chronic gastrointestinal diseases.
4. Diseases found to show clinical significance before screening
5. Combined with diuretics before screening
6. Drugs were used 2 weeks before screening.
7. Laboratory or physical examination with any abnormalities and the researcher's judgment is clinically significant.
8. 12-lead electrocardiogram is abnormal and of clinical significance
9. Positive for hepatitis B surface antigen, positive for hepatitis C antibody, positive for syphilis spirochete antibody, positive for HIV antibody
10. People with severe allergic diseases or known or suspected of being allergic to any of the ingredients in the research drug, allergic constitution (multiple drugs and food allergies)
11. Participated in the clinical trial of any drug or medical device within the first 3 months of screening or planned to participate in the clinical trial of other drugs or medical devices during the trial period (subject to the signing of informed consent)
12. Drink more than 14 units of alcohol per week in the first 6 months of screening; or those who have taken alcohol products 48 hours before administration; or those who have tested positive for alcohol exhalation during the baseline period.
13. Smoking more than 5 cigarettes a day in the 3 months before screening or using any tobacco products 48 h before administration.
14. Drink/eat coffee, tea, grapefruit, chocolate or soft drinks, such as cola containing methamphetrine (tein, caffeine or cocoaine) within 3 days before screening
15. Those who have had a history of drug abuse in the past five years or have used drugs in the first three months of the trial; or urine drugs are screened positive
16. Blood donation ≥ 200 mL within 1 month before screening; or blood donation ≥ 400 mL within 3 months before screening; or trauma or surgical surgery with blood donation (plasma or platelets) or blood loss of ≥ 400 mL within 2 weeks
17. Inability tolerate venous puncture and blood collection or dizziness
18. Subjects who believe that there are other factors that are not suitable to participate in this test

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence and severity of adverse events in healthy subjects after single and multiple doses of HRS-1780 tablets | About a month from the first medication to the evaluation.

SECONDARY OUTCOMES:
Assess the concentration of HRS-1780 in plasma and urine | About 4 weeks after the first dose
Evaluation of AUC0-t of HRS-1780 in plasma and urine | About 4 weeks after the first dose
Evaluation of AUC0-∞ of HRS-1780 in plasma and urine | About 4 weeks after the first dose
Evaluation of Tmax of HRS-1780 in plasma and urine | About 4 weeks after the first dose
Evaluation of Cmax of HRS-1780 in plasma and urine | About 4 weeks after the first dose
Evaluation of t1/2 of HRS-1780 in plasma and urine | About 4 weeks after the first dose
Evaluate the blood pressure of subjects over time after HRS-1780 administration | About 4 weeks after the first dose
Evaluate the heart rate of subjects over time after HRS-1780 administration | About 4 weeks after the first dose
Evaluate the concentrations of plasma renin activity of subjects over time after HRS-1780 administration | About 4 weeks after the first dose
Evaluate the plasma aldosterone of subjects over time after HRS-1780 administration | About 4 weeks after the first dose
Evaluate the plasma angiotensin II of subjects over time after HRS-1780 administration | About 4 weeks after the first dose
Evaluate the urinary creatinine curve of subjects with time after HRS-1780 administration | About 4 weeks after the first dose
Evaluate the change curve of urine creatinine over time relative to baseline in subjects after HRS-1780 administration | About 4 weeks after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shen Q, Li L, Qian W, Dong X, Bao M, Huang R, Li N, Ye Z, Cheng G, Wang Q, Shen K, Luo Z. A four-in-one first-in-human study to assess safety, tolerability, pharmacokinetics, pharmacodynamics, and concentration-QTc relationship of HRS-1780, a selective non-steroidal mineralocorticoid receptor antagonist, in healthy men. Expert Opin Investig Drugs. 2024 Oct;33(10):1083-1093. doi: 10.1080/13543784.2024.2393867. Epub 2024 Aug 26. PMID 39155700